CLINICAL TRIAL: NCT05133687
Title: The Hemodynamic Effects of Different Volumes of Bupivacaine 0.25% Caudal Blocks in Pediatrics Undergoing Lower Abdominal Surgeries as Measured by Electrical Cardiometry: A Randomized Controlled Study
Brief Title: The Hemodynamic Effects of Different Volumes of Bupivacaine 0.25% Caudal Blocks in Pediatrics Undergoing Lower Abdominal Surgeries as Measured by Electrical Cardiometry
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator,Lecturer of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MS-445-2021
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia, Caudal; Pediatrics
Keywords: pediatrics; caudal anesthesia; hemodynamics; electrical cardiometry; bupivacaine 0.25%
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Children will be recruited into the trial during pre-operative assessment. Recruited children will be randomly assigned to one of three groups in a 1:1:1 ratio; (Group 0.8-G) to receive general anesthesia and caudal block with 0.8 ml/kg of bupivacaine 0.25% and (Group 1.2-G) to receive general anesthesia and caudal block with 1.2 ml/kg of bupivacaine 0.25% and (Group G) to receive general anesthesia with local infiltration of the wound or transversus abdominis plan block (TAPB) at the end of the procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The concealed envelopes will be opened by an anesthesia resident (who will not be involved in patient management) and he will be responsible for preparing and giving the caudal block for the caudal groups as instructed in the envelope. the data will be collected by another anesthetist who is blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (0.8-G) (Experimental): This group will receive general anesthesia and caudal block with 0.8 ml/kg of bupivacaine 0.25%
  Interventions: Drug: Bupivacaine Hydrochloride
- Group (1.2-G) (Experimental): This group will receive general anesthesia and caudal block with 1.2 ml/kg of bupivacaine 0.25%
  Interventions: Drug: Bupivacaine Hydrochloride
- Group G (Active Comparator): This group will receive general anesthesia with local infiltration of the wound or transversus abdominis plan block (TAPB) at the end of the procedure.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Recruited children will be randomly assigned to one of three groups in a 1:1:1 ratio; (Group 0.8-G), (Group 1.2-G) and (Group G).

SUMMARY:
This randomized, controlled study is designed to estimate the effects of different volumes of plain bupivacaine 0.25% caudal block on different hemodynamic parameters assessed by electrical cardiometry.

DETAILED DESCRIPTION:
Introduction:

Caudal block is one of the most used regional blocks in pediatrics because it is safe and provides efficient and adequate perioperative analgesia for most of the infra-umbilical and lower limb procedures.[1,2] It has been proposed that the cardiovascular effects of neuraxial blocks are less marked in children than in adults because of lower systemic vascular resistance (SVR) in pediatric population.[3] There is a wide range of doses used in caudal block depending on the desired dermatomal level which can range from 0.5ml/kg up to 1.25ml/kg. [1] However, studies assessing effects and safety of different volumes of caudal blocks on different hemodynamic variables are scarce and show conflicting results due to small sample sizes, absence of control groups, retrospective nature, different additives and different methods for measuring the hemodynamics.[4-8] Electrical Cardiometry (EC) estimates cardiac parameters by measuring changes in thoracic electrical bioimpedance during the cardiac cycle using skin electrodes. It has emerged as a new noninvasive tool for assessment of cardiac output with a good accuracy in adult and pediatric anesthesia.[9] The current study is designed to estimate the effects of different volumes of bupivacaine 0.25% caudal block on different hemodynamic parameters assessed by electrical cardiometry.

Hypothesis:

We hypothesized that different volumes of plain bupivacaine 0.25% caudal block could have direct effects on different hemodynamic parameters in pediatrics undergoing lower abdominal surgeries.

Methods:

The study is a double blinded randomized controlled trial that will be conducted at Abu Al Reesh Children's Hospital, Faculty of Medicine, Cairo University after approval of research and ethics committees.

Children will be recruited into the trial during pre-operative assessment. Recruited children will be randomly assigned to one of three groups in a 1:1:1 ratio; (Group 0.8-G) to receive general anesthesia and caudal block with 0.8 ml/kg of bupivacaine 0.25% and (Group 1.2-G) to receive general anesthesia and caudal block with 1.2 ml/kg of bupivacaine 0.25% and (Group G) to receive general anesthesia with local infiltration of the wound or transversus abdominis plan block (TAPB) at the end of the procedure.

Randomization will be achieved using a computer-generated sequence. Concealment will be achieved using opaque envelopes.

All children will be anesthetized in accordance with the local policy of pediatric anesthesia unit in Abu El-Reesh pediatric hospital-Cairo university.

After preoperative examination and upon arrival to the operating room heart rate HR, noninvasive blood pressure NBP and oxygen saturation SPO2 will be monitored using standard monitor (drȁger infinity vista XL) before inhalational induction of anesthesia using titration of sevoflurane in oxygen air mixture 60% (starting from 3% up to 8%) until the child is put to sleep. Electrical cardiometry device (ICON; Cardiotonic, Osypka; Berlin, Germany) will be applied to the patient through 4 ECG electrodes at the following sites: (forehead, left side of the neck, left mid-axillary line at the level of xiphoid process and left thigh). Patient's sex, height, and weight will be entered into the device, which is set to estimate cardiovascular parameters at a 20-beat moving average recorded every10 seconds. The ECG electrodes will be placed before induction for cooperative children. Baseline electrical cardiometry (ICON) data (Cardiac output, Cardiac index, Stroke volume, Stroke volume variation, Stroke index, Systemic vascular resistance, Systemic vascular resistance index, ICON, VIC, Thoracic fluid index, Left cardiac work, Systolic time ratio, Pre ejection period, Left ventricular ejection time) will be recorded by averaging 3 sets of data over 30 seconds by an anesthesia resident who is blinded to the children groups.

After securing an intravenous line anesthesia will be completed with 1-2µg/kg of fentanyl and atracurium 0.5 mg/kg to facilitate endotracheal intubation. Anesthesia will be maintained by using 1-1.5% isoflurane in a mixture of oxygen and air (50/50) and atracurium top ups at a dose of 0.1mg/kg every 30 minutes.

The concealed envelopes will then be opened by a second anesthesia resident (who will not be involved in patient management) and he will be responsible for preparing and giving the caudal block for the caudal groups as instructed in the envelope.

Children in groups (0.8-G) and (1.2-G) will then be positioned on their right side, and a 22-gauge needle will be aseptically inserted into the caudal epidural space. Bupivacaine 0.25% at a dose of 0.8 ml/kg and 1.2 ml/kg making sure not to exceed a maximum of 2.5 mg/kg will be slowly injected. After repositioning the children on their backs, a 10-min steady-state period without surgical stimulation will be permitted during which a multiple set of measurements will be obtained every 2 minutes (a single set of measurements will be recorded by averaging 3 sets of data over 30 seconds), and surgery will be started after this period. Caudal success will be defined as change of hemodynamics (heart rate and or blood pressure) < 20% of base line parameters to surgical incision without need for additional analgesics or increase of inhalational anesthetics. Patients with caudal failure will be excluded from the study.

In group G the surgery will be started after 10 minutes from the induction of anesthesia where a multiple sets of ICON measurements will be obtained every 2 minutes (a single set of measurements will be recorded by averaging 3 sets of data over 30 seconds), from the previous baseline measurements.

In all groups ICON measurements will be obtained every 10 minutes after start of surgery till the end of surgery.

In all groups HR, NBP, SPO2 and end tidal CO2 will be measured every 2 minutes for 10 minutes after induction of anesthesia then every 10 minutes till the end of surgery.

All children will receive a loading dose of 10 ml/kg of lactated ringer solution over 10 minutes after induction of anesthesia and will be maintained on 3 ml/kg/h lactated ringer solution.

ELIGIBILITY:
Inclusion Criteria:

* All pediatrics ASA I&II aged 1-8 years undergoing elective lower abdominal surgeries.

Exclusion Criteria:

ASA ≥ III. Parents refusal of caudal block. Patients with coagulation disorders (Platelets ≤ 50,000 and/or INR> 1.5). Patients with suspected or proved allergic to local anesthetics. Rash or signs of infection at the injection site. Patients requiring emergency or laparoscopic procedures.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
The percentage of change from the baseline measurement of the cardiac index CI 10 minutes after successful caudal block. | 10 minutes after caudal block.

SECONDARY OUTCOMES:
Electrical cardiometry cardiac index | 30 minutes
mean ABP | 1-2 hours
Incidence of complications: block failure, bradycardia (HR < 80/min) , hypotension (blood pressure <20% of base line) and local anesthesia systemic toxicity (LAST) | 1-2 hours
heart rate | 1-2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided